CLINICAL TRIAL: NCT06548867
Title: Retrospective Analysis of Patients With Metastatic Renal Cell Carcinoma Treated With CABOzantinib: a GENomic Signature for Describing Long-lasting Response
Brief Title: Retrospective Analysis of Patients With Metastatic Renal Cell Carcinoma Treated With CABOzantinib
Acronym: CABOGEN
Status: Recruiting | Type: Observational
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Yghea (Unknown); Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: GOIRC-08-2018
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; Genomic signature; long lasting response; cabozantinib treatment
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: long-lasting responders: Patient long-lasting responders (PFS ≥9 months) to cabozantinib
  Interventions: Drug: Cabozantinib
- Group B: primary refractories: Patient progressed from the start to cabozantinib therapy within 3 months
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Patients must have been treated with cabozantinib after one or more previous therapies for mRCC, as per clinical practise.

SUMMARY:
CABOGEN is a Observational, retrospective, multicenter study that will enroll patients with metastatic clear cell renal carcinoma (mccRCC) treated with cabozantinib after one or more previous lines of treatment that included TKIs, immune checkpoint inhibitors or mTOR inhibitors.

DETAILED DESCRIPTION:
The aim of this study is to describe the genomic profiling of patients with metastatic renal cell carcinoma (mRCC) who are long-lasting responders to treatment with cabozantinib and patients who are not long-lasting responders to the cabozantinib treatment.

The study plan to enroll about 80 patients in 10 Italian centers:

Group A: 40 patients defined as long-lasting responders (PFS ≥ 9 months) Group B: 40 patients defined as primary refractories to cabozantinib (PFS ≤ 3 months)

Tissue samples from nephrectomy or from a metastatic site will be used to perform genomic profiling not older than 5 years.Tissue should be formalin-fixed, paraffin-embedded (FFPE).

Genomic profiling will be performed with a hybrid capture-based next-generation sequencing assay (FoundationONE). The sample will be assayed for all coding exons of 324 cancer-related genes plus select introns from 34 genes that are frequently rearranged in cancer. Sequencing will be performed to a mean exon coverage depth of >500X. The resulting sequences will be analyzed for all classes of genomic alteration, including short variant alterations, copy number alterations, and selected gene fusions or rearrangements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with histological diagnosis of predominantly clear cell carcinoma
* Availability of the tumor tissue from the primary tumor and/or a metastatic site for the genomic profiling analysis not older than 5 years.
* Evaluable disease according to RECIST criteria v 1.1
* Treatment with cabozantinib after one or more previous therapies for mRCC
* Patient progressed from the start to cabozantinib therapy within 3 months or after 9 months
* Any prognosis group according to the IMDC risk score
* Signed informed consent must be obtained for living patients. Patients who died and patient untraceable will be analyzed based on the Authorization no. 9/2016 of the Italian Data Protector Supervisor.

Exclusion Criteria:

* Non-availability of tumor tissue from the primary tumor or a metastatic site for biomarker analysis
* Patient progressed between 3 and 9 months from the beginning of treatment with cabozantinib.
* Non-availability of clinical information useful to evaluate the IMDC risk group at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic clear cell renal carcinoma (mRCC) who are long-lasting responders to treatment with cabozantinib and patients who are not long-lasting responders to the cabozantinib treatment. Cabozantinib treatment receive after one or more previuos therapy for mRCC
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Genomic profiling | 12 months
  to describe genomic profiling of patients with mRCC who are long-lasting responders (PFS ≥9 months) to cabozantinib and describe genomic profiling of patients with rapid disease progression following cabozntinib therapy (PFS≤ 3 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | 12 months
  to describe OS based according to detected genomic profiling
Overall response rate (ORR) | 12 months
  to describe ORR according to the detected genomic profiling
Duration of response (DOR) | 12 months
  to describe duration of response (DOR) according to the detected genomic profilingto describe the genomic profiling according to treatment line (second, third or subsequent) to describe anamnestic characteristics (weight, ECOG PS, sites of metastasis, response to previous treatment lines)

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — AUSL/IRCCS of Reggio Emilia; Cristina Masini, MD, Study Chair — AUSL/IRCCS of Reggio Emilia; Stefania Di Girolamo, MD, Study Chair — AUSL/IRCCS of Reggio Emilia
Locations (1):
- AUSL-IRCCS of Reggio Emilia, Reggio Emilia, Italy